CLINICAL TRIAL: NCT01488487
Title: Phase II Single Arm Study of Everolimus and Pasireotide (SOM230) in Patients With Advanced or Metastatic Hepatocellular Carcinoma (HCC)
Brief Title: Everolimus and Pasireotide (SOM230) in Patients With Advanced or Metastatic Hepatocellular Carcinoma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: UNC Lineberger Comprehensive Cancer Center (Other)
Collaborators: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: LCCC 1032
Record Dates: First submitted 2011-12-06; First posted 2011-12-08 (Estimated); Results first posted 2016-04-07 (Estimated); Last update posted 2016-04-07 (Estimated); Status verified 2016-03

CONDITIONS: Advanced Adult Hepatocellular Carcinoma
Keywords: HCC; Advanced Hepatocellular Carcinoma; Metastatic Hepatocellular Carcinoma; Liver Cancer
MeSH Terms: conditions — Carcinoma, Hepatocellular; Liver Neoplasms | interventions — Everolimus; pasireotide

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Everolimus + pasireotide (Experimental): Oral Everolimus 7.5 mg administered daily for 28 days per cycle, plus pasireotide Long Acting Release (LAR) 60 mg administered by intramuscular injection once per 28 day cycle on day 1.
  Interventions: Drug: Everolimus; Drug: Pasireotide

INTERVENTIONS:
Drug: Everolimus — Everolimus 7.5 mg administered daily for 28 days per cycle until disease progression or unacceptable toxicity.
  Other Names: Afinitor; RAD001
Drug: Pasireotide — Monthly (every 28 days) intramuscular injection of long-acting pasireotide (pasireotide LAR 60 mg) repeated on day 1 of every 28 day cycle until disease progression or unacceptable toxicity.
  Other Names: SOM230; Pasireotide LAR; Pasireotide s.c.

SUMMARY:
The purpose of this study is to estimate the time to disease progression when everolimus and pasireotide are given together in patients with advanced or metastatic HCC who have not had any prior systemic therapy.

DETAILED DESCRIPTION:
This open label, single-arm Phase II study will assess time to progression (TTP) and safety of everolimus and pasireotide in patients with advanced or metastatic hepatocellular carcinoma (HCC) and limited prior systemic therapy. Should this regimen demonstrate efficacy, this will support a Phase III randomized clinical trial of this combination therapy. At least 30 patients will be enrolled into this Phase II study. Additionally, given the potential importance of the RAS/RAF/MEK/ERK and RAS/pAKT pathways, we propose to correlate outcomes with baseline pAKT, p-S6, somatostatin receptor tumor expression, and serum VEGF expression. We anticipate these exploratory analyses will increase understanding of the molecular pathways and their inhibition in this disease. The study will be performed as a University of North Carolina-coordinated, multicenter study.

ELIGIBILITY:
Inclusion Criteria:

* Each subject must meet all of the following inclusion criteria to participate in this study:

  1. Advanced or metastatic hepatocellular carcinoma (stage C per the BCLC criteria, see Appendix A). HCC may be diagnosed by tissue diagnosis or Alpha-fetoprotein (AFP) >400 ng/mL with compatible mass on Magnetic Resonance Imaging Scan (MRI). Cat Scan (CT) abdomen with 3-phase contrast with arterial phase enhancement is acceptable, although MRI is preferred (imaging should be done within 4 weeks of study initiation). Recurrences of previously resected HCC will not require tissue confirmation if there is clear radiographic recurrence in the judgment of the investigator. Disease must not otherwise be amenable to local therapy.
  2. Maximum Childs-Pugh score 6 (see Appendix A) with no active encephalopathy
  3. Prior systemic therapy limited to sorafenib that was discontinued due to intolerance. Patients must undergo at least a 4-week washout prior to enrollment.
  4. Eastern Cooperative Oncology Group (ECOG) PS of 0-2
  5. Life expectancy of >12 weeks
  6. Age ≥18 years
  7. Patients who have received previous local therapy, such as surgery, radiotherapy, hepatic arterial embolization, chemoembolization, radiofrequency ablation, percutaneous injection, or cryoablation, will be eligible for enrollment in the study provided that there is documented progression and disease is not amenable to further local therapies. Therapy must be completed >4 weeks prior to study initiation (Day 1 of everolimus and pasireotide administration).
  8. Minimum of 4 weeks since any major surgery
  9. No active serious infection or other comorbid illness which would impair ability to participate in the trial.
  10. International Normalized Ratio (INR) ≤1.5. (Anticoagulation is allowed if target INR ≤2.0 on a stable dose of warfarin or on a stable dose of low molecular weight heparin (LMWH) for >2 weeks at time of enrollment).
  11. Fasting serum cholesterol ≤300 mg/dL OR ≤7.75 mmol/L AND fasting triglycerides (TGs) ≤2.5 x upper limit of normal (ULN). NOTE: In case one or both of these thresholds are exceeded, the patient can only be included after initiation of appropriate lipid lowering medication.
  12. Patients must have adequate organ function as evidenced by:

      * Absolute neutrophil count (ANC) ≥1.5 x 109/L
      * Platelet count ≥50 x 109/L
      * Hemoglobin (Hg) >9 g/dL
      * Bilirubin ≤2 x ULN
      * Aspartate transaminase (AST) or Alanine transaminase (ALT) ≤5 x ULN
      * Serum creatinine ≤1.5 x ULN OR creatinine clearance ≥50 mL/min (estimated by Cockcroft Gault or measured)
  13. Serum magnesium and serum potassium within institutional normal limits (patients may be on replacement)
  14. Women of childbearing potential (WOCBP) must have a negative serum or urine pregnancy test performed within 7 days prior to Day 1 of everolimus and pasireotide administration.
  15. WOCBP and men must agree to use adequate contraception (barrier method of birth control) prior to study entry and for the duration of study participation. Men and women should use adequate birth control for at least 8 weeks after the last administration of study drugs. (Oral, implantable, or injectable contraceptives may be affected by cytochrome P450 interactions and are therefore not considered effective for this study.)
  16. Signed, Institutional Review Board (IRB) approved written informed consent

Exclusion Criteria:

* Patients meeting any of the following exclusion criteria at baseline will be excluded from study participation:

  1. Patients who have received prior treatment with an mTOR inhibitor (e.g., sirolimus, temsirolimus, everolimus) or somatostatin analog (e.g. octeotride)
  2. Chronic treatment with systemic steroids (except for intermittent topical, local injection, or eye drops) or another immunosuppressive agent. NOTE: This restriction regarding systemic steroids does not apply should patient need course of glucocorticoid for treatment of non-infectious pneumonitis during study (see Section 4.5.2).
  3. Patients with a known hypersensitivity to everolimus or other rapamycins (e.g., sirolimus, temsirolimus) or to its excipients
  4. Patients with a known hypersensitivity to somatostatin or to its excipients
  5. Concurrent or planned radiation, hormonal, chemotherapeutic, experimental, or targeted biologic therapy
  6. Prior treatment with any investigational drug within the preceding 4 weeks
  7. Patients who have any severe and/or uncontrolled medical conditions or other conditions that could affect their participation in the study such as:

     * Symptomatic congestive heart failure (New York Heart Association [NYHA] Class III or IV)
     * Unstable angina pectoris, symptomatic congestive heart failure, myocardial infarction within 6 months of start of study drug, serious uncontrolled cardiac arrhythmia, or any other clinically significant cardiac disease
     * Severely impaired lung function as defined as spirometry and diffusing capacity for carbon monoxide (DLCO) that is 50% of the normal predicted value and/or 02 saturation that is 88% or less at rest on room air
     * Uncontrolled diabetes as defined by fasting serum glucose >1.5 x ULN or Glycated hemoglobin (HbA1c) >8.0% (Note: at the principle investigator's discretion, ineligible patients can be re-screened after adequate medical therapy has been instituted.)
     * Active (acute or chronic) or uncontrolled severe infections. NOTE: A detailed assessment of Hepatitis B/C medical history and risk factors must be done at screening for all patients. Hepatitis B viral deoxyribonucleic acid (HBV DNA) and Hepatitis C viral ribonucleic acid (HCV RNA) polymerase chain reaction (PCR) testing are required at screening for all patients with a positive medical history based on risk factors and/or confirmation of prior HBV/HCV infection. See Section 4.2 for further information.
  8. Clinically significant third space fluid accumulation (i.e., ascites requiring paracentesis despite use of diuretics) or pleural effusion that either requires thoracentesis or is associated with shortness of breath
  9. Risk factors for prolongation of Corrected QT Interval (QTc)* including:

     * QTc at screening >450 msec
     * History of syncope or family history of idiopathic sudden death
     * Sustained or clinically significant cardiac arrhythmias
     * Risk factors for Torsades de Pointes such as hypokalemia, hypomagnesemia, cardiac failure, clinically significant/symptomatic bradycardia, or high-grade AV block
     * Concomitant disease(s) that could prolong QT such as autonomic neuropathy (caused by diabetes or Parkinson's disease), human immunodeficiency virus (HIV), uncontrolled hypothyroidism, or cardiac failure
     * Concomitant medication(s) known to increase QT interval (See Appendix B)

       * University of North Carolina at Chapel Hill (UNC) uses GE electrocardiogram (ECG) carts which use the Bazett formula for QTc.
  10. Patients should not receive immunization with attenuated live vaccines within 1 week of study entry or during study period. Close contact with those who have received attenuated live vaccines should be avoided during treatment with everolimus. Examples of live vaccines include intranasal influenza, measles, mumps, rubella, oral polio, Bacillus Calmette-Guérin (BCG), yellow fever, varicella, and TY21a typhoid vaccines.
  11. Uncontrolled brain or leptomeningeal metastases, including patients who continue to require glucocorticoids for brain or leptomeningeal metastases
  12. Symptomatic cholelithiasis
  13. Other malignancies within the past 3 years except for adequately treated carcinoma of the cervix or basal or squamous cell carcinomas of the skin
  14. A known history of HIV seropositivity (HIV testing is not mandatory)
  15. Impairment of gastrointestinal function or gastrointestinal disease that may significantly alter the absorption of everolimus (e.g., ulcerative disease, uncontrolled nausea, vomiting, diarrhea, malabsorption syndrome, or small bowel resection.)
  16. Patients with an active, bleeding diathesis or on oral anti-vitamin K medication (except warfarin as long as the goal INR is ≤1.5). Low-molecular-weight heparin (LMWH) is permitted (see Section 3.1.10.)
  17. Unable or unwilling to discontinue use of prohibited fruit (or its juices) and/or prohibited medications listed in Appendix B for at least 14 days or five half-lives of a drug (whichever is longer) prior to the first dose of study drug and for the duration of the study
  18. Male patient whose sexual partner(s) are WOCBP who are not willing to use adequate contraception during the study and for 8 weeks after the end of treatment
  19. Active alcohol intake of 80 grams or more per day. For reference, one portion of alcohol (one glass of wine, one can or bottle of beer, or one ounce of hard liquor) contains approximately 15 grams of ethanol.
  20. Inability to comply with study and/or follow-up procedures
  21. History of noncompliance to medical regimens

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2011-12; Primary Completion 2015-03 (Actual); Study Completion 2015-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Hanna Sanoff, MD, Principal Investigator — University of North Carolina at Chapel Hill Lineberger Comprehensive Cancer Center
Locations (3):
- United States (3):
  - Moffitt Cancer Center, Tampa, Florida
  - University of North Carolina at Chapel Hill Lineberger Comprehensive Cancer Center, Chapel Hill, North Carolina
  - Comprehensive Cancer Center of Wake Forest University, Winston-Salem, North Carolina

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: UNC Lineberger Website — http://unclineberger.org

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Of the 33 participants screened for eligibility, 24 were deemed eligible and went on to treatment, 8 were ineligible, and 1 participant withdrew consent prior to treatment assignment.
Groups:
- Everolimus + Pasireotide: Oral Everolimus 7.5 mg administered daily for 28 days per cycle, plus pasireotide LAR 60 mg administered by intramuscular injection once per 28 day cycle on day 1.
  Everolimus: Everolimus 7.5 mg administered daily for 28 days per cycle until disease progression or unacceptable toxicity.
  Pasireotide: Monthly (every 28 days) intramuscular injection of long-acting pasireotide (pasireotide LAR 60 mg) repeated on day 1 of every 28 day cycle until disease progression or unacceptable toxicity.
Period: Overall Study
Arm/Group | Everolimus + Pasireotide
Started | 24
Received Treatment | 24
Completed | 15
Not Completed | 9
Not completed — Adverse Event | 6
Not completed — Death | 1
Not completed — Withdrawal by Subject | 2

BASELINE CHARACTERISTICS:
Population: Patients assigned to treatment
Arm/Group | Everolimus + Pasireotide
Number analyzed (Participants) | 24
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 15
  >=65 years | 9
Age, Continuous [Median (Full Range); unit: years] | 59 [23 to 87]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8
  Male | 16
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 24
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 2
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 1
  White | 21
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 24
Chronic Hepatitis C [Number; unit: participants] — Presence of Hepatitis C virus as a cause of hepatocellular carcinoma
  participants
    Present | 7
    Absent | 17
Chronic Hepatitis B [Number; unit: participants] — Presence of Hepatitis B virus as a cause of hepatocellular carcinoma
  participants
    Present | 2
    Absent | 22
Child-Pugh Score (Stage) [Median (Full Range); unit: units on a scale] — A scale to assess severity of liver disease based on five clinical features: 1) serum bilirubin, 2) serum albumin, 3) prothrombin time, 4) the degree of ascites, and 5) the grade of hepatic encephalopathy. One point given for absent/normal, 2 points for slight or mild, and 3 points for severe. Child-Pugh Score could range from 5 - 15, with lower scores equaling better prognosis.
  units on a scale | 5 [5 to 6]
Time from diagnosis to enrollment [Median (Full Range); unit: Months] | 4 [1 to 88]
CLIP (Cancer of the Liver Italian Program) score [Median (Full Range); unit: units on a scale] — The CLIP score for a patient with hepatocellular carcinoma is calculated by assigning a score (0, 1 or 2) to each of four clinical factors: a) Child-Pugh stage; b) number of tumor nodules and whether the tumor extends through <=50% or >50% of the liver; c) AFP; and d) portal vein thrombosis.
  These scores are added together to yield a CLIP score of 0-6, with lower scores having a better outcome.
  units on a scale | 1.5 [0 to 5]
BCLC (Barcelona Clinic Liver Cancer) Stage [Number; unit: participants] — Missing for one participant. Barcelona Clinic Liver Cancer (BCLC) staging criteria ranges from very early stage (0), to early stage (A), Intermediate stage (B), advanced stage (C), and end stage (D). Staging is based on Child-Pugh score, performance status, and number and size of nodules. Earlier stages (0,A) have better prognosis.
  participants
    Stage B | 2
    Stage C | 21
    Missing | 1
Portal vein involvement [Number; unit: participants]
  Present | 9
  Absent | 15
Extent of cancer [Number; unit: participants]
  Unifocal | 2
  Multifocal | 11
  Metastatic | 11
Prior therapy received for this cancer [Number; unit: participants receiving this prior tx] — Participants may have received more than one type of prior therapy.
  participants receiving this prior tx
    Transarterial chemoembolization (TACE) | 4
    Transarterial radioembolization (TARE) | 2
    Ablation | 2
    Surgery | 8
    None | 12
    Missing | 1

OUTCOME MEASURES:

1. Primary Outcome: Time to Progression (TTP)
Description: Time to progression is defined as the time from study enrollment until radiological progression in a previously embolized lobe, development of new lesions in an untreated lobe, or evidence of extrahepatic progression (based on modified Hepatocellular Carcinoma (HCC) Response Evaluation Criteria In Solid Tumors (RECIST) criteria). Patients will be followed until death. Patients that die of causes unrelated to the study drug without evidence of progression will be censored.
Time Frame: 3.5 years
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Everolimus + Pasireotide
Number analyzed (Participants) | 24
months | 3.5 [2 to 5.8]

2. Secondary Outcome: Number of Individuals Experiencing Toxicity
Description: Safety determinations are based on the rate of drug-related adverse events (AEs) reported based upon the toxicity as measured by the NCI Common Terminology Criteria for Adverse Events version 4.0 (CTCAE v4.0).
Time Frame: 3.5 years
Measure: Number; unit: participants
Arm/Group | Everolimus + Pasireotide
Number analyzed (Participants) | 24
participants
  Dose Limiting Toxicities (DLT) | 1
  Any adverse event | 24

3. Secondary Outcome: Overall Survival (OS)
Description: Overall survival is defined as the time from study enrollment until death.
Time Frame: 3.5 years
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Everolimus + Pasireotide
Number analyzed (Participants) | 24
months | 6.7 [6 to NA] — The upper limit of the 95% Confidence Interval was calculated as infinity (and thus NA) due to few events at the time of analysis.

4. Secondary Outcome: Objective Response Rate (ORR)
Description: ORR is the rate of complete responses (CRs) + partial responses (PRs) as determined by RECIST (v1.1) and modified HCC RECIST criteria. Responses defined as follows:
  CR: disappearance of all clinical/radiological evidence of tumor including any intratumoral arterial enhancement in all target lesions.
  Partial Response (PR): at least a 30% decrease in the sum of diameters of viable (contrast enhancement in the arterial phase) target lesions, referencing the baseline sum.
  Stable Disease (SD): any cases that do not qualify for either partial response or progressive disease.
  Progressive Disease (PD): an increase of at least 20% in the sum of the diameters of viable target lesions, referencing the nadir sum, and/or the appearance of one or more new lesions. A new hepatic nodule signals PD when the longest diameter is at least 10 mm and the nodule shows the typical vascular pattern of HCC on dynamic imaging or if at least 1-cm interval growth is seen in subsequent scans.
Time Frame: 3.5 years
Population: Two patients were not evaluable; one due to death prior to radiographic evaluation (death clinically attributed to progressive disease) and the other due to early termination of treatment due to intolerance.
Measure: Number; unit: percentage of participants
Arm/Group | Everolimus + Pasireotide
Number analyzed (Participants) | 22
percentage of participants
  Radiographic response (CR or PR) | 0
  Stable disease | 45.5

ADVERSE EVENTS:
Time Frame: Followed for 4 weeks after treatment
Arm/Group | Everolimus + Pasireotide
Serious Adverse Events (participants affected / at risk) | 6/24
Other Adverse Events (participants affected / at risk) | 24/24
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Everolimus + Pasireotide (N=24)
Stroke (Nervous system disorders) | 2 (2) — Unlikely to be related to treatment
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Confusion (Psychiatric disorders) | 1 (2)
Death NOS (General disorders) | 2 (2) — Death within 30 days of treatment; related to disease, not treatment
Diarrhea (Gastrointestinal disorders) | 1 (1)
Dizziness (Nervous system disorders) | 1 (1)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Fatigue (General disorders) | 1 (1)
Generalized Muscle Weakness (Musculoskeletal and connective tissue disorders) | 2 (3)
Hepatobiliary Disorders - Other, Specify (Hepatobiliary disorders) | 1 (1) — Hepatic Failure
Hypokalemia (Metabolism and nutrition disorders) | 2 (2)
Mucositis Oral (Gastrointestinal disorders) | 1 (1)
Pleural Effusion (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Rectal Hemorrhage (Gastrointestinal disorders) | 1 (1)
Weight Loss (Investigations) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 4% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Everolimus + Pasireotide (N=24)
Abdominal Pain (Gastrointestinal disorders) | 2 (3)
Activated Partial Thromboplastin Time Prolonged (Investigations) | 1 (1)
Alanine Aminotransferase Increased (Investigations) | 10 (11)
Alkaline Phosphatase Increased (Investigations) | 10 (14)
Anemia (Blood and lymphatic system disorders) | 8 (8)
Anorexia (Metabolism and nutrition disorders) | 3 (3)
Aspartate Aminotransferase Increased (Investigations) | 13 (16)
Back Pain (Musculoskeletal and connective tissue disorders) | 2 (2)
Blood Bilirubin Increased (Investigations) | 5 (8)
Chest Pain - Cardiac (Cardiac disorders) | 1 (1)
Cholesterol High (Investigations) | 3 (3)
Confusion (Psychiatric disorders) | 2 (2)
Constipation (Gastrointestinal disorders) | 2 (2)
Cough (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Diarrhea (Gastrointestinal disorders) | 9 (10)
Dysgeusia (Nervous system disorders) | 1 (1)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Edema Limbs (General disorders) | 1 (1)
Fatigue (General disorders) | 7 (8)
Fever (General disorders) | 1 (1)
Flu Like Symptoms (General disorders) | 1 (1)
Hemoglobin Increased (Investigations) | 1 (1)
Hyperglycemia (Metabolism and nutrition disorders) | 16 (50)
Hypertension (Vascular disorders) | 1 (1)
Hypertriglyceridemia (Metabolism and nutrition disorders) | 4 (4)
Hypocalcemia (Metabolism and nutrition disorders) | 1 (1)
Hypomagnesemia (Metabolism and nutrition disorders) | 1 (1)
Hypophosphatemia (Metabolism and nutrition disorders) | 1 (2)
Hypotension (Vascular disorders) | 1 (1)
Insomnia (Psychiatric disorders) | 1 (1)
Lower Gastrointestinal Hemorrhage (Gastrointestinal disorders) | 1 (1)
Lymphocyte Count Decreased (Investigations) | 1 (2)
Mucositis Oral (Gastrointestinal disorders) | 8 (10)
Muscle Weakness Upper Limb (Musculoskeletal and connective tissue disorders) | 1 (1)
Nausea (Gastrointestinal disorders) | 3 (5)
Nervous System Disorders - Other, Specify (Nervous system disorders) | 1 (1) — Encephalopathy Confusion
Neutrophil Count Decreased (Investigations) | 3 (3)
Pain (General disorders) | 2 (4)
Pain In Extremity (Musculoskeletal and connective tissue disorders) | 1 (1)
Palmar-Plantar Erythrodysesthesia Syndrome (Skin and subcutaneous tissue disorders) | 1 (1)
Platelet Count Decreased (Investigations) | 6 (8)
Pruritus (Skin and subcutaneous tissue disorders) | 1 (1)
Rash Acneiform (Skin and subcutaneous tissue disorders) | 1 (1)
Rash Maculo-Papular (Skin and subcutaneous tissue disorders) | 5 (6)
Rectal Hemorrhage (Gastrointestinal disorders) | 1 (1)
Stomach Pain (Gastrointestinal disorders) | 1 (1)
Vomiting (Gastrointestinal disorders) | 3 (3)
Weight Loss (Investigations) | 1 (1)
White Blood Cell Decreased (Investigations) | 2 (3)

LIMITATIONS AND CAVEATS:
Unplanned interim analysis due to negative results from another trial found conditional probability of rejecting null hypothesis based on events in the 24 patients enrolled was 0.08. Accrual goals had been met and study was complete per protocol.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes